CLINICAL TRIAL: NCT03680235
Title: Novel Intervention to Increase Lactation Practices by African American Women
Brief Title: Informational Intervention in Increasing Lactation Practices by African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I 270615; NCI-2018-00854 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 270615 (Other: Roswell Park Cancer Institute); R21CA202263 (NIH)
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subject; Pregnant
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I: (standard information about pregnancy, breastfeeding) (Active Comparator): Participants receive standard information about pregnancy and breastfeeding. Participants may also participate in a focus group with their partner/spouse or family members after the baby's birth.
  Interventions: Other: Informational Intervention; Other: Interview; Other: Survey Administration
- Group II (information about breastfeeding and cancer) (Experimental): Participants receive standard information about pregnancy and breastfeeding as well as information about breastfeeding and breast cancer. Participants may also participate in a focus group with their partner/spouse or family members after the baby's birth.
  Interventions: Other: Informational Intervention; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Receive standard information about breastfeeding and pregnancy
Other: Informational Intervention — Receive information about breastfeeding and cancer
  Arms: Group II (information about breastfeeding and cancer)
Other: Interview — Participate in focus groups
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies how well an informational intervention works in increasing lactation practices by African American women. Giving additional information about breastfeeding and breast cancer risks to African American women may help doctors understand the factors that affect the decision to breast feed and to test whether providing useful information about breastfeeding will change breastfeeding behavior.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop appropriate intervention strategies about the "breastfeeding-breast cancer connection" appropriate for use by experienced Women, Infants and Children (WIC) Peer Counselors (PCs) to disseminate to African-American mothers through a community-based participatory research (CBPR) approach including social media..

II. Assess the comparative cognitive (e.g., knowledge, utility, cost-benefit), affective association (e.g., feelings), socioeconomic, familial and intent/outcome (e.g., breastfeeding) measures pre- and post-intervention to determine effectiveness of the content to impact cognitive and feeling measures and increase breastfeeding in young African-American mothers compared to an existing counseling program.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I: Participants receive standard information about pregnancy and breastfeeding. Participants may also participate in a focus group with their partner/spouse or family members after the baby's birth.

GROUP II: Participants receive standard information about pregnancy and breastfeeding as well as information about breastfeeding and breast cancer. Participants may also participate in a focus group with their partner/spouse or family members after the baby's birth.

After completion of the information intervention, participants are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant African American women participating in the Catholic Charities WIC Program
* INCLUSION - FOCUS GROUPS: Representative mothers, spouses/partners, influential family members (e.g., grandmothers, sisters) from the families served during the study.
* INCLUSION - FOCUS GROUPS: Partners/spouses may include men or women.

Exclusion Criteria:

* Unwilling or unable to follow protocol requirements.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding rates | Up to 1 year
  Will be assessed by estimating a logistic regression model with breastfeeding as the dichotomous outcome variable and intervention condition as a predictor variable.
Behavioral intentions for breastfeeding | Up to 1 year
  Linear regression analyses will be conducted with condition and necessary covariates as predictors.
Perceived risk for breast cancer | Up to 1 year
  Linear regression analyses will be conducted with condition and necessary covariates as predictors. Will examine the degree to which perceived risk for breast cancer mediate any intervention impact on breastfeeding behavior and behavioral intentions.
Affective associations with breastfeeding | Up to 1 year
  Linear regression analyses will be conducted with condition and necessary covariates as predictors. Will examine the degree to which affective associations with breastfeeding mediate any intervention impact on breastfeeding behavior and behavioral intentions.
Perceptions of benefits and barriers to breastfeeding | Up to 1 year
  Linear regression analyses will be conducted with condition and necessary covariates as predictors. Will examine the degree to which perceptions of benefits and barriers to breastfeeding mediate any intervention impact on breastfeeding behavior and behavioral intentions.
Qualitative analysis of focus group and key informant interviews | Up to 1 year
  Will be recorded and transcribed. This text will be coded and categorized by Erwin following methods established in earlier research. The PEN-3 Model analysis will focus on the most salient factors as they apply to what will be considered the ?Positive, Existential, Negative? influences within the Cultural Empowerment domain in reference to breastfeeding and formula feeding topics. Will sort the responses into categories in a 3 x 3 table according to the Relationships and Expectations domain factors, ?Perceptions, Enablers, Nurturers,? on one axis, and the ?Positive, Existential, Negative? factors across the other axis. This categorical analysis will be reviewed and edited and the Women, Infants and Children (WIC) peer counselors (PCs) to increase validity of the process.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Erwin, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Dauphin C, Clark N, Cadzow R, Saad-Harfouche F, Rodriguez E, Glaser K, Kiviniemi M, Keller M, Erwin D. #BlackBreastsMatter: Process Evaluation of Recruitment and Engagement of Pregnant African American Women for a Social Media Intervention Study to Increase Breastfeeding. J Med Internet Res. 2020 Aug 10;22(8):e16239. doi: 10.2196/16239. PMID 32773377